CLINICAL TRIAL: NCT06704620
Title: Safety and Effectiveness of Tislelizumab and Platinum-based Chemotherapy Combination With H1 Receptor Antagonist（Diphenhydramine）in Advanced and Metastatic Non-Small Cell Lung Cancer: A Prospective, Randomized-controlled, Multi-center, Open-label, Phase-III Trial.
Brief Title: Study of Tislelizumab and Platinum-based Chemotherapy Combination With H1 Receptor Antagonist（Diphenhydramine）in Advanced and Metastatic Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241045
Record Dates: First submitted 2024-11-12; First posted 2024-11-26 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Advanced and Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Diphenhydramine; tislelizumab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1 (Experimental): Tislelizumab intravenous infusion 200mg d1; Pemetrexed intravenous infusion 500mg/m2 d1 or Albumin paclitaxel intravenous infusion 260mg/m2 d1; Carboplatin intravenous infusion AUC5 d1 or Cisplatin intravenous infusion 75mg/m2 d1; Diphenhydramine intramuscular injection 20mg qd d0-2 Q3W
  Interventions: Drug: Diphenhydramine; Drug: Tislelizumab; Drug: Pemetrexed; Drug: Albumin paclitaxel; Drug: Carboplatin; Drug: Cisplatin
- Arm2 (Active Comparator): Tislelizumab intravenous infusion 200mg d1; Pemetrexed intravenous infusion 500mg/m2 d1 or Albumin paclitaxel intravenous infusion 260mg/m2 d1; Carboplatin intravenous infusion AUC5 d1 or Cisplatin intravenous infusion 75mg/m2 d1; Q3W
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed; Drug: Albumin paclitaxel; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Diphenhydramine — Diphenhydramine intramuscular injection 20mg qd d0-2 Q3W
  Arms: Arm1
Drug: Tislelizumab — Tislelizumab intravenous infusion 200mg d1
Drug: Pemetrexed — Pemetrexed intravenous infusion 500mg/m2 d1
Drug: Albumin paclitaxel — Albumin paclitaxel intravenous infusion 260mg/m2 d1
Drug: Carboplatin — Carboplatin intravenous infusion AUC5 d1
Drug: Cisplatin — Cisplatin intravenous infusion 75mg/m2 d1

SUMMARY:
The goal of this clinical trial is to learn if diphenhydramine can improve the effectiveness and decrease the toxicity for the treatment of advanced and metastatic Non-small cell lung cancer (NSCLC) with PD1 inhibitor plus chemotherapy.

The main questions it aims to answer are:

* Dose diphenhydramine improve the effectiveness and survival of advanced and metastatic NSCLC treated with PD1 inhibitor and chemotherapy?
* Dose diphenhydramine decrease the toxicity of PD1 inhibitor plus platinum-based chemotherapy?
* Researchers will compare patients with or without diphenhydramine to see if diphenhydramine works to improve the effectiveness and decrease the toxicity.

Participants will:

* Take standard treatment (tislelizumab and platinum-based chemotherapy) with/without diphenhydramine（20mg qd d0-2）every cycle.
* Visit the clinic once every six weeks for checkups and tests
* Keep a diary of their symptoms and survival visit based on the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent before implementing any procedures related to the trial;
2. Age ≥18 years old and ≤75 years old;
3. ECOG score 0 or 1;
4. Expected survival time >3 months;
5. Patients diagnosed with stage IIIB-IV NSCLC by imaging, tissue and/or cytology (according to AJCC 9th edition), or primary stage IIIB-IV NSCLC that relapses after surgery (if adjuvant therapy has been used, the drug must be discontinued for more than 6 months);Patients with IIIB/C are unable to undergo radical surgery or radiotherapy; Patients (adenocarcinoma and adenosquamous carcinoma) with wide type EGFR and negative ALK fusion gene can enroll into the trial;
6. Not received systemic antitumor therapy before;
7. Included patients were intended to receive Tirellizumab combined with standard chemotherapy containing platinum. Squamous lung cancer patients should use Paclitarel for Injee in(Albumin Bound) plus platinum, non-squamous patients should use pemetrexed plus platinum;
8. There was at least one radiographically measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST version 1.1). Lesions located within the field of previous radiotherapy may be considered measurable if progression is demonstrated.
9. The subject is allowed to receive palliative radiation therapy (including craniocerebral radiation therapy for symptomatic brain metastases) and radiation-related toxicities recover to less than or equal to degree 1(CTCAE 5.0, except hair loss).
10. For adequate organ function, the subject must meet the following laboratory criteria:

1) The absolute value of neutrophil (ANC) ≥1.5x109/L in the past 14 days without the use of granulocyte colony-stimulating factor; 2) Platelets ≥100×109/L without blood transfusion in the past 14 days; 3) Hemoglobin >9g/dL in the last 14 days without blood transfusion or use of erythropoietin; 4) Total bilirubin ≤1.5 times the upper limit of normal (ULN) 5) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) in ≤2.5 times ULN (subject with liver metastasis allowed ALT or AST ≤5×ULN); 6) Serum creatinine ≤1.5 times ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min; 7) Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; 8) Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is out of normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can also be enrolled; 9) Myocardial enzyme profiles within the normal range (laboratory abnormalities that are not clinically significant as determined by the investigator) are also allowed); 11. For female subjects of childbearing age, they should be administered for urine or blood pregnancy tests and the results should be negative within 3 days prior to the first study drug administration (day 1 of cycle 1). If the urine pregnancy test results cannot be confirmed as negative, blood pregnancy tests is required. Women of non-childbearing age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy; 12. If there is a risk of pregnancy, all subjects (male or female) are required to take contraception with an annual failure rate of less than 1% was within 120 days after drug administration (or 180 days after last study drug administration) in the study for the entire duration of treatment until the end of treatment

Exclusion Criteria:

1. Patients with lung metastasis of other primary malignant tumors;
2. Patients with previous or concurrent malignant tumors of other systems (excluding basal cell carcinoma of skin and squamous dermatocarcinoma after radical treatment. and/or carcinoma in situ after radical resection);
3. Patients received perioperative immunotherapy (preoperative neoadjuvant or postoperative adjuvant);
4. With known driver gene mutations such as EGFR/ALK/ROS1;
5. Patients with existing or previously diagnosed myasthenia gravis;
6. Patients with existing or previously diagnosed angle-closure glaucoma;
7. Patients with existing or previously diagnosed prostatic hypertrophy;
8. Patients were allergic to diphenhydramine and its excipients;
9. Patients with pyloric-duodenal obstruction, pyloric stenosis caused by peptic ulcer, and bladder neck stenosis;
10. Received radiation therapy prior to administration of the drug in the first study, meeting one of the following conditions:

1) ≥30% of bone marrow had received radiation therapy within 14 days prior to treatment 2) Received radiation therapy for lung lesions within 6 weeks prior to treatment with a dose >30Gy (Enrolled subjects must be safe from the toxicity of prior radiation therapy (Recover to grade 1 or below), no need for glucocorticoid therapy and no history of radiation pneumonia) 11. Patients are currently participating in an interventional clinical study treatment or has received another investigational drug or used research instrument therapy within 4 weeks prior to initial dosing.

12. Received proprietary Chinese medicines with anti-cancer indications or immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural fluid) systemic treatment; 13. Patients have had active autoimmune diseases occurred within 2 years prior to first administration agents, which need for systemic treatment (e.g. use of disease-modifying drugs, glucocorticoids, or immunosuppression). Alternative therapies (e.g., thyroxine, insulin or for adrenal or pituitary machines) Incomplete physiological glucocorticoids, etc.) are not considered as systemic treatment; 14. Systemic glucocorticoid therapy (excluding nasal, inhalation, or other means for local use) was being received within 7 days prior to the first administration of the study) or any other form of immunosuppressive therapy; Note: Physiological doses of glucocorticoids are permitted (≤10 mg/ day of prednisone or equivalent); 15. There is clinically uncontrollable pleural effusion/abdominal effusion (Subjects no need to drain the effusion or no significant increase in effusion after 3 days of stopping drainage can be enrolled); 16. Known allogeneic organ transplantation (other than corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 17. The patient has not fully recovered from the toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or in baseline, excluding weakness or hair loss); 18. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 19. Untreated active hepatitis B (defined as HBsAg positive with a detectable HBV-DNA copy number greater than upper limit of normal value in cardiac laboratory);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load <1000 copies /ml (200 IU/ml) prior to initial dosing, subjects should be treated with chemotherapy drugs throughout the study during this period, anti-HBV therapy is taken to avoid viral reactivation
2. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-), no need to receive prophylactic anti-HBV therapy, but close monitoring of viral reactivation is required.

20. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection); 21. Received live vaccine within 30 days prior to the first dose (cycle 1, day 1); Note: Injectable inactivated virus vaccine against seasonal influenza is permitted for 30 days prior to initial administration; But it is not allowed to receive intranasal live attenuated flu vaccine.

22. Pregnant or lactating women; 23. The presence of any serious or uncontrolled systemic disease, such as:

1. There is a significant abnormality in the rhythm, conduction or morphology of the resting electrocardiogram with severe symptoms that are difficult to control, such as the complete left bundle branch conduction block, heart block above degree II, ventricular arrhythmia or atrial fibrillation;
2. Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure;
3. Myocardial infarction occurred within 6 months before enrollment;
4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
5. There is a history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to initial administration, or there is a current clinical activity interstitial lung disease;
6. Active pulmonary tuberculosis;
7. There is an active or uncontrolled infection that requires systemic treatment;
8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
11. Urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0 g;
12. Subjects with mental disorders who are unable to cooperate with treatment; 24. Medical history or evidence of disease, treatment, or laboratory tests that may interfere with the test results or prevent the subject from participating fully in the study. The investigator considered the subjects with other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 24 months
  From the initial treatment until the date of disease progression or the date of death from any cause, whichever occurred first

SECONDARY OUTCOMES:
ORR | up to 24 months
  ORR was defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR)
OS | 3 years
  OS was the time from the initial treatment until the date of death from any cause
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events[Safety and Tolerability] | up to 24 months
  Adverse events were assessed according to the National Cancer Insti- tute Common Terminology Criteria for Adverse Events, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Liu, M.D,Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No